CLINICAL TRIAL: NCT01812239
Title: Vaginal Progesterone to Prevent Early Preterm Birth In Twin Pregnancy With Short Cervix. Double-Blind, Placebo-Controlled, Randomized Clinical Trial
Brief Title: Vaginal Progesterone in Twins With Short Cervix
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: inability to retain study drug with comparable placebo.
Sponsor: Obstetrix Medical Group (Industry)
Responsible Party: Sponsor
Organization: Pediatrix (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OBX0019
Record Dates: First submitted 2013-03-12; First posted 2013-03-18 (Estimated); Last update posted 2014-12-19 (Estimated); Status verified 2014-12

CONDITIONS: Premature Birth
Keywords: premature birth; twins; short cervix
MeSH Terms: conditions — Premature Birth | interventions — Progestins; Fibronectins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vaginal Progesterone (Active Comparator): Daily administration of Vaginal Progesterone (200mg) Gel between 20 weeks of pregnancy and 34 weeks of pregnancy.
  Interventions: Drug: Vaginal Progesterone gel.; Procedure: fetal fibronectin swab.
- Placebo (Placebo Comparator): Daily vaginal administration of Placebo gel (Vanicream)between 20 weeks of pregnancy and 34 weeks of pregnancy.
  Interventions: Procedure: fetal fibronectin swab.; Drug: Placebo gel

INTERVENTIONS:
Drug: Vaginal Progesterone gel. — Daily administration of Vaginal Progesterone gel in pregnant women with twins between the 20th week of pregnancy and the 34th week of pregnancy.
  Other Names: progestin
  Arms: Vaginal Progesterone
Procedure: fetal fibronectin swab. — Collection of quantatative fetal fibronectin swab one week after randomization into the trial for both arms. Randomziation occurs between 20 weeks - 24 weeks of gestation.
  Other Names: fFN; fibronectin
Drug: Placebo gel — weekly vaginal administration of the placebo gel from randomization until 34 weeks of gestation.
  Other Names: placebo
  Arms: Placebo

SUMMARY:
A Multicenter, Double-Blind, Placebo-Controlled Randomized Clinical Trial of Vaginal Progesterone to Prevent Early Preterm Birth In Twin Pregnancy with Short Cervix.

DETAILED DESCRIPTION:
This is a placebo-controlled, double-blind, randomized clinical trial of asymptomatic women with twin pregnancy and a cervix length 10 mm to 25 mm discovered on a routine screening transvaginal sonogram between 20w0d to 24w0d gestational age. Women will be randomized in either the in-patient or out-patient setting (1:1) to a daily vaginal application of micronized progesterone cream(200 mg)vs. placebo to determine if daily vaginal progesterone administration reduces the risk of preterm birth prior to 34w0d of gestation.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age between 20w0d and 24w0d
* Twin pregnancy, diamniotic-dichorionic, both twins living
* Cervical length 10 mm to 25 mm discovered by a screening transvaginal ultrasound exam

Exclusion Criteria:

* Mother less than 18 years of age
* Uterine contractions of 40 seconds duration or more, 10 or more per hour
* Rupture of fetal membranes (leakage of amniotic fluid one or both sacs)
* Ongoing vaginal bleeding
* Any condition likely to cause serious neonatal morbidity independent of gestational age, including:

  1. fetal malformation likely to require surgery
  2. fetal malformation involving vital organs
  3. fetal viral infection
  4. hydrops fetalis
  5. discordance in estimated fetal weight more than 10%
  6. velamentous insertion of umbilical cord of either twin
  7. placenta previa of either placenta
* Any contraindication to continuing the pregnancy
* Cervical cerclage in place or planned
* Any contraindication to vaginal micronized progesterone, including:

  1. Known sensitivity to progesterone or any of the other ingredients
  2. Liver dysfunction or disease
  3. Known or suspected malignancy of breast or genital organs
  4. Active thromboembolic disorder, or history of hormone-associated thromboembolic disorder

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2014-03; Primary Completion 2017-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Birth of baby before 34 weeks of gestation | At the time of delivery
  The primary outcome is defined as Early Preterm Birth, that is, birth before 34weeks of gestation. A birth at 33weeks 6days or earlier is considered to have the primary outcome. A birth at 34weeks 0days or later does not have the primary outcome. Births for any reason before 34weeks 0days are considered to have the primary outcome, whether they are "spontaneous" or not.

SECONDARY OUTCOMES:
Gestational age of baby at birth | measure at time of birth
  measured of the average Gestational age of babies at birth.
Rate of "spontaneous birth" before 34weeks of gestation | from randomization to birth of the baby - up to 15 weeks
  Rate of "spontaneous birth" before 34weeks of gestation. Spontaneous births are those whose underlying cause is judged to be due to preterm labor, prelabor rupture of membranes, or cervical insufficiency. (In contradistinction, "indicated" deliveries are those due to preeclampsia, fetal growth problems, fetal heart rate abnormalities, and other problems.)
Rate of composite neonatal morbidity | measures from randomization to 60 days post delivery of the baby
  Composite morbidity is defined as any one or more of: stillbirth, neonatal death, infant death before hospital discharge, respiratory distress syndrome (RDS), intracranial hemorrhage (grade 3 or 4)(IVH), necrotizing enterocolitis (stage 2 or 3)(NEC), documented neonatal sepsis within 72 hr of birth, or periventricular leukomalacia (characteristic lesions in the subcortical white matter seen on cerebral imaging studies within 96 hrs of birth)(PVL).

OTHER OUTCOMES:
Comparison of effectiveness of progesterone in women in highest 2 quartiles of quantitative fetal fibronectin (fFN) versus those in the lowest 2 quartiles of quantitative fFN. | from the 21st week of gestation until the 25 week of gestation
  A cervicovaginal swab for quantitative fetal fibronectin testing will be obtained at the first antenatal visit, approximately 1 week after enrollment. The results of this will be used to test a secondary hypothesis that fFN levels will identify a subgroup of participants who respond to progesterone treatment and another subgroup who do not.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Combs, MD, Principal Investigator — Pediatrix
Locations (1):
- Good Samaritan Hospital, San Jose, California, United States